CLINICAL TRIAL: NCT06617949
Title: Evaluating Pain Control Strategies in Postpartum Patients on Opioid Use Disorder Medications: Efficacy and Safety Outcomes.
Brief Title: Evaluating Pain Control Strategies in Postpartum Patients on Opioid Use Disorder Medications.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Christopher Fadumiye, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00052798
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Substance Use Disorder (SUD)
Keywords: Pain conrtrol; Substance use disorder; Parturient
MeSH Terms: conditions — Substance-Related Disorders | interventions — Anesthesia, Conduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Transverse abdominal Plane(TAP) Block with long acting Exparel (Active Comparator): A subset of participants (n=15) will be divided into three different arms: A.) Postoperative Epidural infusion for 24-36hrs B.) Hydromorphone Patient Controlled Analgesia (PCA) with Preservative free Morphine via epidural for 36hrs C.) Transverse abdominal Plane(TAP) Block with long acting Exparel.
  Interventions: Drug: Regional Anesthesia
- Postoperative Epidural infusion for 24-36hrs (Active Comparator): A subset of participants (n=15) will be divided into three different arms: A.) Postoperative Epidural infusion for 24-36hrs B.) Hydromorphone Patient Controlled Analgesia (PCA) with Preservative free Morphine via epidural for 36hrs C.) Transverse abdominal Plane(TAP) Block with long acting Exparel.
  Interventions: Procedure: Epidural local anesthetic infusion
- Hydromorphone Patient Controlled Analgesia (PCA),Preservative free Morphine via epidural for 36hrs (Active Comparator): A subset of participants (n=15) will be divided into three different arms: A.) Postoperative Epidural infusion for 24-36hrs B.) Hydromorphone Patient Controlled Analgesia (PCA) with Preservative free Morphine via epidural for 36hrs C.) Transverse abdominal Plane(TAP) Block with long acting Exparel.
  Interventions: Drug: Hydromorphone Patient Controlled Analgelsic

INTERVENTIONS:
Drug: Regional Anesthesia — Transverse abdominal Plane(TAP) Block with long acting Exparel placed by a regional anesthesiologist.
  Arms: Transverse abdominal Plane(TAP) Block with long acting Exparel
Drug: Hydromorphone Patient Controlled Analgelsic — This group will be administered epidural PCA as a modality for pain control post cesarian section
  Arms: Hydromorphone Patient Controlled Analgesia (PCA),Preservative free Morphine via epidural for 36hrs
Procedure: Epidural local anesthetic infusion — Epidural group will receive pain control via a local anesthetic intermediate bolus infusion
  Arms: Postoperative Epidural infusion for 24-36hrs

SUMMARY:
The purpose of this study is to investigate the efficacy of three different modalities of post-operative pain control in parturient with opioid use disorders. The investigators aim to determine whether the different approach utilized show better outcomes with pain management and if there are any association with reduction of symptoms of anxiety, depression, and overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include being a parturient with Substance use disorder (SUD) and age 18-35

Exclusion Criteria:

* Exclusion criteria include having a diagnosed medical condition(allergies to medication, pathology such as severe aortic stenosis excluding patients from receiving an epidural etc) that will exempt patient from intervention arm of the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Change in pain assessment scores from baseline post surgery | immediately after the study intervention and up to post op day 2
  Number of participants with significant change in pain assessment scores and any association with reduction of symptoms of anxiety, depression, and overall well-being.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Froedtert Hospital Milwaukee, Wisconsin 53226, Milwaukee, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data, statistical analysis and conclusions.
Supporting Information: Study Protocol, SAP